

## **Results Summary**

# Protocol Title: Cranial electric stimulation (CES) to modify suicide risk factors in psychiatric inpatients

**Study No.:** HP-00065640, Date January 4th 2018

Principal Investigator: Nithin Krishna MD, 410-328-6610, 410-328-5386 (24 hour access)

ClinicalTrials.gov Identifier: NCT02846740

Christopher E. Stamper and Christopher A. Lowry Statisticians.

### **Data Preprocessing:**

Random forest analysis does not support missing values. The following experimental variables were removed prior to analysis because there were more than 2 missing values.

HAMAT1, HAMAT2, MADRA\_T2, MADRA\_T3, PSQI\_T2, PSQI\_T3, T2time, compositetotalT2, granulocytespercent, granulocyteabsolute, lymphocyteabsloute, lymphocytepercent, monocyteabsolute, monocytepercent, basophileabs, basophiperc, eosinophilabd, Eosinphilsperc, nucleatedrbcabs, nucleatedrbcperc, MCH, MCHC, Immaturegransabs, Immaturegranspec, Magnesium, Phosphorus, TotalProtein, Albumin, AST, ALT, TotalBilirubin, AlkPhos, TSH, VITB12, Folate

If the number of missing values in an experimental variable was less than or equal to 2 the value was changed to the median of the column and documented below.

The following data points were altered:

Level of confidence for participant CES005 was changed from blank to 3 (the median of the column). This was the only missing value in this column.

wbc for participant CES030 was changed from blank to 7.8 (the median of the column). This was the only missing value in this column.

hb for participant CES030 was changed from blank to 13 (the median of the column). This was the only missing value in this column.

htc for participant CES030 was changed from blank to 40.1 (the median of the column). This was the only missing value in this column.

platelets for participant CES030 was changed from blank to 285 (the median of the column). This was the only missing value in this column.

MCV for participant CES030 was changed from blank to 87.2 (the median of the column). This was the only missing value in this column.

MPV for participant CES019 and CES030 was changed from blank to 9.85 (the median of the column). These were the only missing values in this column.

RDW for participant CES030 was changed from blank to 13.6 (the median of the column). This was the only missing value in this column.

Sodium for participant CES019 and CES030 was changed from blank to 139 (the median of the column). These were the only missing values in this column.

Potassium for participant CES019 and CES030 was changed from blank to 3.95 (the median of the column). These were the only missing values in this column.

Chloride for participant CES030 was changed from blank to 104 (the median of the column). This was the only missing value in this column.

CO2 for participant CES019 and CES030 was changed from blank to 27 (the median of the column). These were the only missing values in this column.

AnionGap for participant CES019 and CES030 was changed from blank to 9 (the median of the column). These were the only missing values in this column.

BUN for participant CES019 and CES030 was changed from blank to 12.5 (the median of the column). These were the only missing values in this column.

Creatinine for participant CES019 and CES030 was changed from blank to .785 (the median of the column). These were the only missing values in this column.

Glucose for participant CES019 and CES030 was changed from blank to 94 (the median of the column). These were the only missing values in this column.

Calcium for participant CES019 and CES030 was changed from blank to 9 (the median of the column). These were the only missing values in this column.

The following experimental variables were removed because the values were identical to the treatment codes. Actual\_Devise\_Used\_ACTIVE\_vs.\_Sham

The following experimental variables were added to examine the change between the last observation and the baseline observation for the primary target variables.

MADRA\_Delta: MADRALAST\_OBS – MADRA\_Baseline\_T0 HAMAT\_Delta: HAMLAST\_OBS – HAMAT0 PSQI\_Delta: PSQILAST\_OB – PSQI\_T1

See the attached csv file, "Alpha stim data" for the data that were used in the analysis.

#### Method

Analysis done in R Version 3.4.1

### **Random forest results:**

All random forest models were run to create 2001 trees.

Random forest model predicting treatment group (Active vs Sham)

OOB (out-of-bag) error rate: 60%

• This means that the model was wrong 60% of the time and correct 40% of the time.

Here is a plot showing how the model is converging as the number of trees increases. Overall this is the inverse of what you would want to see. Optimally you want the error to start high and decrease to a convergence or a plateau as the number of trees increases. The convergence is settling at an error of  $\sim$ 0.6, which is your OOB error rate.



For reference this is what a more favorable plot looks like. This plot has an OOB error rate of 5.73%.



Back to your data, here are the experimental variables that are most predictive of treatment group. There are 2 accuracy metrics here that are used interchangeably based on the preference of the investigator. The accuracy numbers are a bit arbitrary and there is no threshold of significance per se. These are simply the most predictive variables of the target experimental variable.

rf



Random forest model predicting Montgomery-Asberg Depression Scale change between the final observation and baseline (MADRA Delta)

The MADRA\_Delta score is continuous; therefore, the model produces a % variation explained rather than an OOB error rate.

% variation explained: 14.14%

• Meaning that ~85% of the variation is unexplained

Here is the plot showing how the model is converging. Again the model is not converging very well.



Here are the experimental variables that are explaining the most variation or are the most predictive of the MADRA\_Delta score. It is encouraging that HAMAT\_Delta score and PSQI-Delta score are two of the best predictors of MADRA\_Delta score.



rf

Page 5 of 15

 $Random\ forest\ model\ predicting\ Hamilton\ Depression\ Score\ change\ between\ the\ final\ observation\ and\ baseline\ (HAMAT\_Delta)$ 

% variation explained: 0.83%

## • Meaning that ~99% of the variation is unexplained

Here is the plot showing how the model is converging. Again the model is not converging very well.



Here are the experimental variables that are explaining the most variation or are the most predictive of the HAMAT\_Delta score. It is encouraging that MADRA\_Delta score is one of the best predictors of HAMAT\_Delta score.



Random forest model predicting Pittsburg Sleep Quality Index score change between the final observation and baseline (PSQI Delta).

% variation explained: 13.01%

## • Meaning that ~87% of the variation is unexplained

Here is the plot showing how the model is converging. Better.





Random forest model predicting Length of Stay (LOS).

% variation explained: 18.7%

• Meaning that ~81% of the variation is unexplained

Here is the plot showing how the model is converging.



Here are the experimental variables that are explaining the most variation or are the most predictive of the LOS.

rf



I made some box plots of the target variables with notches. If the notches are overlapping that means that the difference is not significant.

# MADRA\_Delta



# HAMAT\_Delta







I also ran some linear models on the target variables to see if there was a significant proportion of the variation explained by the treatment. Here are the various models. A summary of the results is that none of the target variables explained a significant proportion of the variance in the treatment variable. In addition the treatment variable did not explain a significant proportion of the variance in any of the target variables.

#### Active vs Sham

```
Call:
lm(formula = dat$Active_vs._Sham ~ dat$MADRA_Delta + dat$PSQI_Delta +
   dat$LOS + dat$HAMAT_Delta)
Residuals:
   Min
           1Q Median
                          30
                                Max
-0.7116 -0.4783 0.1233 0.4296 0.6952
Coefficients:
               Estimate Std. Error t value Pr(>|t|)
(Intercept)
              dat$MADRA_Delta -0.008970 0.014086 -0.637
                                           0.530
dat$PSQI_Delta 0.024970 0.021857 1.142
                                           0.264
dat$LOS
              -0.014567
                        0.011225 -1.298
                                           0.206
dat$HAMAT_Delta 0.006887
                        0.019592 0.352
                                          0.728
Signif. codes: 0 '*** 0.001 '** 0.01 '* 0.05 '.' 0.1 ' 1
Residual standard error: 0.5104 on 25 degrees of freedom
Multiple R-squared: 0.1317, Adjusted R-squared: -0.007216
F-statistic: 0.9481 on 4 and 25 DF, p-value: 0.4529
```

MADRA Delta

```
Call:
lm(formula = dat$MADRA_Delta ~ dat$HAMAT_Delta + dat$PSQI_Delta +
   dat$Active_vs._Sham + dat$LOS)
Residuals:
    Min
              1Q Median
                               30
                                       Max
                           4.8098 13.4379
-19.1440 -4.4362
                   0.3207
Coefficients:
                    Estimate Std. Error t value Pr(>|t|)
(Intercept)
                    -4.75714
                               4.17875 -1.138 0.265741
dat$HAMAT_Delta
                    0.84571
                               0.21889 3.864 0.000703 ***
                               0.28752 2.271 0.032044 *
dat$PSQI_Delta
                    0.65285
dat$Active_vs._Sham1 -1.77929
                               2.79430 -0.637 0.530071
dat$LOS
                    -0.07574
                               0.16263 -0.466 0.645431
___
Signif. codes: 0 '*** 0.001 '** 0.01 '* 0.05 '.' 0.1 ' ' 1
Residual standard error: 7.188 on 25 degrees of freedom
Multiple R-squared: 0.5498, Adjusted R-squared: 0.4778
F-statistic: 7.633 on 4 and 25 DF, p-value: 0.0003661
```

 $HAMAT\_Delta$ 

```
Call:
lm(formula = dat$HAMAT_Delta ~ dat$MADRA_Delta + dat$PSQI_Delta +
    dat$Active_vs._Sham + dat$LOS)
Residuals:
    Min
              1Q
                   Median
                               3Q
                                       Max
-10.2459 -2.5605 0.1305 1.8374 11.9851
Coefficients:
                    Estimate Std. Error t value Pr(>|t|)
(Intercept)
                    -5.84565
                               2.86952 -2.037 0.052353 .
dat$MADRA_Delta
                    0.44207
                               0.11442 3.864 0.000703 ***
                              0.22805 -0.239 0.812978
dat$PSQI_Delta
                   -0.05453
dat$Active_vs._Sham1 0.71411
                              2.03158 0.352 0.728154
dat$LOS
                    0.26534
                              0.10549 2.515 0.018688 *
Signif. codes: 0 '*** 0.001 '** 0.01 '* 0.05 '.' 0.1 ' '1
Residual standard error: 5.197 on 25 degrees of freedom
Multiple R-squared: 0.5646, Adjusted R-squared: 0.4949
F-statistic: 8.104 on 4 and 25 DF, p-value: 0.000247
```

PSQI Delta

```
Call:
lm(formula = dat$PSQI_Delta ~ dat$MADRA_Delta + dat$HAMAT_Delta +
    dat$Active_vs._Sham + dat$LOS)
Residuals:
               10
     Min
                     Median
                                  30
                                          Max
-11.3494 -2.1282
                     0.1626
                              1.9709
                                       9.8305
Coefficients:
                      Estimate Std. Error t value Pr(>|t|)
                       0.65390
                                  2.71122
                                            0.241
                                                      0.811
(Intercept)
dat$MADRA_Delta
                      0.26188
                                  0.11534
                                            2.271
                                                      0.032 *
dat$HAMAT_Delta
                      -0.04184
                                  0.17500 -0.239
                                                      0.813
dat$Active_vs._Sham1 1.98695
                                  1.73926 1.142
                                                     0.264
dat$LOS
                                  0.10311 -0.406
                      -0.04182
                                                     0.688
Signif. codes: 0 '*** 0.001 '** 0.01 '* 0.05 '.' 0.1 ' ' 1
Residual standard error: 4.553 on 25 degrees of freedom
Multiple R-squared: 0.2684,
                                 Adjusted R-squared: 0.1513
F-statistic: 2.293 on 4 and 25 DF, p-value: 0.08759
LOS
Call:
lm(formula = dat$LOS ~ dat$MADRA_Delta + dat$PSOI_Delta + dat$Active_vs._Sham +
   dat$HAMAT_Delta)
Residuals:
           1Q Median
   Min
                         30
                               Max
-12.844 -4.353 -2.341 2.845 23.249
Coefficients:
                  Estimate Std. Error t value Pr(>|t|)
                             3.3876 5.916 3.57e-06 ***
(Intercept)
                   20.0404
dat$MADRA_Delta
                   -0.1136
                             0.2438 -0.466 0.6454
                             0.3854 -0.406
dat$PSQI_Delta
                   -0.1563
                                            0.6885
dat$Active_vs._Sham1 -4.3329
                             3.3387 -1.298
                                            0.2062
dat$HAMAT_Delta
                   0.7611
                             0.3026
                                     2.515 0.0187 *
Signif. codes: 0 '***' 0.001 '**' 0.01 '*' 0.05 '.' 0.1 ' ' 1
Residual standard error: 8.802 on 25 degrees of freedom
Multiple R-squared: 0.3168,
                            Adjusted R-squared: 0.2075
F-statistic: 2.898 on 4 and 25 DF, p-value: 0.04239
```